CLINICAL TRIAL: NCT06566261
Title: A Phase 1 Open-label, Single Ascending Dose Study of ABA-101 in Participants With Progressive Multiple Sclerosis
Brief Title: ABA-101 in Participants With Progressive Multiple Sclerosis
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Abata Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 101-PMS-101
Record Dates: First submitted 2024-08-20; First posted 2024-08-22 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-06

CONDITIONS: Progressive Multiple Sclerosis
Keywords: Progressive Multiple Sclerosis; Cell Therapy; Multiple Sclerosis; Treg; Regulatory T Cell
MeSH Terms: conditions — Multiple Sclerosis, Chronic Progressive; Multiple Sclerosis

STUDY DESIGN:
Intervention Model Description: Sequential Escalating Dose Cohorts
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- ABA-101 Dose 1 (Experimental): Low Dose ABA-101
  Interventions: Biological: ABA-101
- ABA-101 Dose 2 (Experimental): High Dose ABA-101
  Interventions: Biological: ABA-101

INTERVENTIONS:
Biological: ABA-101 — ABA-101 is a TCR engineered, autologous regulatory T cell (Treg) therapy

SUMMARY:
This study will test the safety and effects of ABA-101 when given as a single dose to participants with progressive multiple sclerosis.

It is the first study of this treatment in humans. After safety is demonstrated with a low dose of ABA-101, a higher dose will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Is ≥18 years old at signing of consent.
* Has a diagnosis of MS per the 2017 revised McDonald criteria.
* Has documented evidence of progression of disability independent of MS relapse activity (clinical or radiographic).
* Expresses the HLA that matches the TCR restriction.
* Presence of a radiographic biomarker of CNS inflammation as identified by MRI.
* Meets Expanded Disability Status Scale (EDSS) criteria.
* Meets the nine-hole peg test (9HPT) criteria.

Exclusion Criteria:

* Presents with clinical or radiographic evidence of relapse within 24 months prior to or at Screening.
* Is considered by the Investigator to be immunocompromised.
* Current treatment with disease-modifying therapies (DMTs).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2024-09-11 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events (safety and tolerability) | Day of Treatment to End of DLT Evaluation Period (28 Days)
  Incidence of AEs through Day 29

CONTACTS AND LOCATIONS:
Overall Officials: Samantha Singer, President and CEO, Abata Therapeutics, MS MBA, Study Director — Abata Therapeutics
Locations (3):
- United States (3):
  - Johns Hopkins University, Baltimore, Maryland
  - Rutgers, Robert Wood Johnson Medical School, New Brunswick, New Jersey
  - Cleveland Clinic Mellen Center, Cleveland, Ohio

IPD SHARING:
Plan to Share IPD: No